CLINICAL TRIAL: NCT05908682
Title: A Single-arm Safety Study of Subjects Exposed to Ibrexafungerp Whilst Pregnant, Including Infant Outcomes Up to One Year
Brief Title: Safety of Pregnant Subjects Exposed to Ibrexafungerp Including Infant Outcomes
Status: Recruiting | Type: Observational
Sponsor: Scynexis, Inc. (Industry)
Collaborators: AWINSA (Unknown)
Responsible Party: Sponsor
Other Study IDs: SCY-078-401
Record Dates: First submitted 2023-06-08; First posted 2023-06-18 (Actual); Last update posted 2024-07-17 (Actual); Status verified 2024-07

CONDITIONS: Vulvovaginal Candidiasis; Candida Infection; Vaginal Candidiasis
Keywords: VVC; Thrush; BREXAFEMME; Candidiasis; Vaginal Yeast; Yeast Infection
MeSH Terms: conditions — Candidiasis, Vulvovaginal; Candidiasis; Candidiasis, Oral

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Study Cohort: Subjects who have been treated with Brexafemme (Ibrexafungerp) at any time during pregnancy or whose conception is estimated to have occurred within four days after receiving the last dose of Brexafemme.
  Interventions: Other: Non-interventional study

INTERVENTIONS:
Other: Non-interventional study — This is not an interventional study

SUMMARY:
This is an ongoing evaluation of subjects exposed to ibrexafungerp while pregnant. The study population will include pregnant women of any age.

DETAILED DESCRIPTION:
This is a single-arm safety study which comprises an ongoing evaluation of subjects exposed to ibrexafungerp while pregnant. The study population will include pregnant women of any age who were exposed to ibrexafungerp during pregnancy, or whose conception is estimated to have occurred within four days after receiving last dose of ibrexafungerp, and are volunteering to take part in this study. Subjects will be monitored starting from exposure during pregnancy until one year after live delivery.

Information on pregnancy outcomes and complications as well as fetal/neonatal/infant outcomes will be collected during the timeframe described in the protocol.

Subjects can enroll in the study by calling the telephone number directly (1-888-982-7299) or through SCYNEXIS BREXAFEMME Pregnancy Study Webpage, OR her healthcare provider (HCP) can, with her consent, enroll her on her behalf.

Data will be collected both retrospectively and prospectively using a variety of questionnaire that will be completed by the representative based on interview with the subject and/or HCP

ELIGIBILITY:
Inclusion Criteria:

1. Exposure to ibrexafungerp during pregnancy or if conception is estimated to have occurred within 4 days of the last dose of ibrexafungerp
2. Subject and/or parent/legal representative consents to participate and agrees to the conditions and requirements of the study including the interview schedule/completion of questionnaire and release of medical records

   * Subject can be identified by the sponsor or HCP, in terms of confirmed pregnancy.

A self-reported pregnancy will be considered as confirmed pregnancy if the Urine Pregnancy Test (UPT) result is positive.

* A woman can self-enroll in the study or her healthcare provider (HCP), with her consent, can enroll her on her behalf.

Exclusion Criteria:

1. Females who were not exposed to safety study medications during pregnancy
2. Refusal to participate in the study
3. An inability to provide an accurate medical history or give informed consent

Min Age: 0 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The study population will include women who were exposed to ibrexafungerp at any time during pregnancy or whose conception is estimated to have occurred within four days after receiving last dose of ibrexafungerp, volunteering to take part in this study.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-07-28 (Actual); Primary Completion 2029-10-31 (Estimated); Study Completion 2029-10-31 (Estimated)

PRIMARY OUTCOMES:
Major Structural Defects | From Brexafemme exposure up to one year after birth
  To collect and describe selected fetal/neonatal/infant outcomes (i.e., major and minor congenital malformations, small for gestational age, and postnatal growth and development) at birth and through up to the first year of life of infants born to women exposed to ibrexafungerp during the defined pregnancy exposure window

SECONDARY OUTCOMES:
To collect and describe pregnancy outcomes | From Brexafemme exposure up to one year post birth
  Live birth, spontaneous abortions, stillbirths, elective abortions, and preterm births

CONTACTS AND LOCATIONS:
Locations (1):
- AWINSA, New Delhi, Vasant Vihar, India

IPD SHARING:
Plan to Share IPD: No